CLINICAL TRIAL: NCT01391975
Title: A Multi Centre Randomized Controlled Trial of the Clinical and Cost Effectiveness of Duplex Ultrasound Surveillance With Proactive Intervention Versus no Surveillance and Reactive Intervention for the Management of Stenosis in Arterio-venous Fistulae for Dialysis Vascular Access.
Brief Title: Surveillance and Proactive Intervention for Dialysis Access
Acronym: SPIDA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Access 6
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Renal Failure; Arteriovenous Fistula
Keywords: arteriovenous fistula; surveillance; arterial stenosis; venous stenosis
MeSH Terms: conditions — Renal Insufficiency; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surveillance and proactive intervention (Experimental)
  Interventions: Procedure: Active ultrasound surveillance of fistula and proactive treatment of stenosis
- Control and reactive intervention (No Intervention)

INTERVENTIONS:
Procedure: Active ultrasound surveillance of fistula and proactive treatment of stenosis — Regular duplex ultrasound assessment of fistula from time of creation until 6 months post procedure with referral of all haemodynamically significant stenoses to further imaging and treatment
  Arms: Surveillance and proactive intervention

SUMMARY:
Newly formed dialysis fistulae can often fail, and failure is usually due to narrowing of the blood vessels. Methods of detecting narrowing are available and, more importantly, can detect narrowings before a fistula fails. It is not known whether treating these narrowings will actually improve fistula survival or if the majority can be left alone. we wish to see if we can detect such narrowings with ultrasound scanning and if early detection and treatment improves patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Incident patients referred to vascular or transplant surgery departments for primary AV fistula formation for haemodialysis access.
2. Ability to give informed written consent
3. Aged over 18 at time of referral

Exclusion Criteria:

1. Inability to give informed written consent
2. Aged under 18 at time of referral
3. Inability to attend follow-up appointments

Specific exclusion;

1. Previous arteriovenous access procedures in target limb
2. Unsuitable for upper limb radiocephalic or brachiocephalic AVF formation
3. Known thrombophilic or thrombotic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Cumulative or secondary patency | within 6 months of fistula formation
  This being the interval from the time of access placement until access abandonment, thrombosis, or the time of patency measurement including intervening manipulations (surgical or endovascular interventions) designed to re-establish functionality in thrombosed access.

SECONDARY OUTCOMES:
Number of thrombosis events | within 6 months of fistula formation
Number of fistula failures | within 6 months of fistula formation
Number, type and technical success rate for elective interventions | within 6 months of fistula formation
Number, type and technical success rate of acute interventions | within 6 months of fistula formation

CONTACTS AND LOCATIONS:
Locations (1):
- Hull Royal Infirmary, Hull, United Kingdom